CLINICAL TRIAL: NCT00295503
Title: A Phase II Trial of Cisplatin, Pemetrexed and Bevacizumab in Untreated Malignant Mesothelioma
Brief Title: Cisplatin, Pemetrexed and Bevacizumab for Untreated Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: University of Chicago (Other); Columbia University (Other); Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVF3442S
Record Dates: First submitted 2006-02-22; First posted 2006-02-23 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-09

CONDITIONS: Mesothelioma
Keywords: mesothelioma; bevacizumab; chemotherapy
MeSH Terms: conditions — Mesothelioma | interventions — Bevacizumab; Cisplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): cisplatin, pemetrexed, and bevacizumab
  Interventions: Drug: bevacizumab; Drug: cisplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: bevacizumab — 15 mg/kg IV every 3 weeks
Drug: cisplatin — 75 mg/m2 IV every 3 weeks
Drug: pemetrexed — 500 mg/m2 every 3 weeks

SUMMARY:
To estimate the time to progression of cancer in patients with previously untreated mesothelioma receiving cisplatin, pemetrexed and bevacizumab

DETAILED DESCRIPTION:
Secondary endpoints will include:

objective response rate

overall survival

In addition, the objective of the analysis of the correlative science data is to determine any association between tumor expression of VEGF/KDR complex and/or the presence of sv40 (as detected by PCR amplification) and objective response.

ELIGIBILITY:
Inclusion criteria

5.2.1 Patients must have histologically proven malignant mesothelioma (epithelial, sarcomatoid, or mixed subtype) not amenable to curative surgery or radiotherapy. Eligible sites of origin include the pleura, peritoneum, and tunica vaginalis.

5.2.2 Patient's disease must not be amenable to curative treatment with surgery. Evidence of gross unresectability will include but not be limited to direct extension into the chest wall, mediastinal or hilar lymphadenopathy, pulmonary or cardiac function that is inadequate to tolerate resection, and sarcomatoid or mixed histology.

5.2.3 Patients must be > 18 years old 5.2.4 Patients must have measurable disease.

Adequate organ function and functional status

Exclusion Criteria:

a. General Medical Concerns 5.3.1 Patients must not be pregnant or breast feeding. 5.3.2 No "currently active" second malignancy other than non-melanoma skin cancer. Patients are not considered to have a "currently active" second malignancy if they have completed therapy and have a less than 30% risk of relapse.

5.3.3 No uncontrolled intercurrent illness including but not limited to: active infection, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, or psychiatric/social situations that would limit compliance with study requirements.

5.3.4 No HIV positive patients receiving combination anti-retroviral therapy because of possible pharmacokinetic interactions with study medications.

5.3.5 History of allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab or other agents used in the study.

5.3.6 Inability to interrupt aspirin or other non-steroidal medication for a 5 day period.

c. Bevacizumab-Specific Concerns

Subjects meeting any of the following criteria are ineligible for study entry:

5.3.7 Patients with brain metastases are excluded 5.3.8 History of myocardial infarction or CVA (stroke) within 6 months of study entry.

5.3.9 Evidence of bleeding diathesis or coagulopathy. Patients on therapeutic doses of coumadin are eligible as long as the INR is maintained in the range of 2-3 and there is no evidence of active bleeding.

5.3.10 Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study 5.3.11 Urine protein:creatinine ratio less than 1.0 at screening 5.3.12 Serious, non-healing wound, ulcer, or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Dowell, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from investigators clinics
Groups:
- Cisplatin, Pemetrexed and Bevacizumab: cisplatin 75 mg/m2, pemetrexed 500 mg/m2 and bevacizumab 15 mg/kg IV every 3 weeks
Period: Overall Study
Arm/Group | Cisplatin, Pemetrexed and Bevacizumab
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: one patient excluded due to ineligibility. That patient is included in the toxicity analysis
Groups:
- Cisplatin, Pemetrexed and Bevacizumab: cisplatin 75 mg/m2, pemetrexed 500 mg/m2, and bevacizumab 15 mg/kg IV every 3 weeks
Arm/Group | Cisplatin, Pemetrexed and Bevacizumab
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 28
Age, Continuous [Median (Full Range); unit: years] | 66 [24 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 44
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 6 Months
Description: This is the percentage of patients alive and progression-free at 6 months from initiation of treatment.
Time Frame: patients progression free at 6 months
Measure: Number; unit: percentage of participants
Groups:
- Cisplatin, Pemetrexed, Bevacizumab: cisplatin 75 mg/m2, pemetrexed 500 mg/m2 and bevacizumab 15 mg/kg IV every 3 weeks
Arm/Group | Cisplatin, Pemetrexed, Bevacizumab
Number analyzed (Participants) | 52
percentage of participants | 56

2. Secondary Outcome: Response Rate
Description: response was assessed by the RECIST criteria (version 1.0). Per those criteria, progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: from time of enrollment to time of best response or death from any cause, whichever came first up to 100 months
Measure: Number; unit: percentage of participants
Arm/Group | Cisplatin, Pemetrexed, Bevacizumab
Number analyzed (Participants) | 52
percentage of participants | 40

3. Secondary Outcome: Overall Survival
Description: overall survival was measured from time of initiation of treatment to death from any cause
Time Frame: From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up 100 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin, Pemetrexed and Bevacizumab
Number analyzed (Participants) | 52
months | 14.8 [10.0 to 17.0]

ADVERSE EVENTS:
Time Frame: 3 years 6 months
Groups:
- Experimental Arm: cisplatin, pemetrexed, and bevacizumab
Arm/Group | Experimental Arm
Serious Adverse Events (participants affected / at risk) | 16/53
Other Adverse Events (participants affected / at risk) | 24/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=53)
pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 5 (5)
deep venous thrombosis (Vascular disorders) | 3 (3)
RPLS (Nervous system disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1)
small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
neutropenic fever (Blood and lymphatic system disorders) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
squamous cell carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=53)
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — Grade 3/4 neutropenia only
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) — Grade 3 and 4 only
Anemia (Blood and lymphatic system disorders) | 1 (1) — Grade 3 and 4 only
Fatigue (General disorders) | 4 (4) — Grade 3 and 4 only
Constipation (Gastrointestinal disorders) | 2 (2) — Grade 3 and 4 only
Dehydration (General disorders) | 2 (2) — Grade 3 and 4 only
Neuropathy (Nervous system disorders) | 2 (2) — Grade 3 and 4 only
Allergic reaction (Immune system disorders) | 1 (1) — Grade 3 and 4 only
Anorexia (General disorders) | 1 (1) — Grade 3 and 4 only
Creatinine (Renal and urinary disorders) | 1 (1) — Grade 3 and 4 only
Mucositis (Gastrointestinal disorders) | 1 (1) — Grade 3 and 4 only
Vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3 and 4 only

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No